CLINICAL TRIAL: NCT00163371
Title: Effect of Ciclesonide (320 mcg/Day) vs Fluticasone Propionate (375 mcg/Day) vs. Placebo on Short-term Linear Growth Rate and HPA-axis Function in Prepubertal Children With Mild Asthma
Brief Title: Effects of Inhaled Ciclesonide Versus Fluticasone Propionate Versus Placebo on Lower Leg Growth in Prepubertal Children With Mild Persistent Asthma (6 to 12 y) (BY9010/M1-208)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-208
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Child; Fluticasone propionate; HPA-axis; Pediatric; Linear growth rate
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to compare the effects of ciclesonide inhaled at one dose level twice daily versus fluticasone propionate inhaled at one dose level twice daily versus placebo, on short-term lower leg growth in prepubertal children with mild persistent asthma. The study duration consists of a baseline period (2 weeks), a treatment period (2 weeks for each treatment), and a wash-out period (2 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent by the patient's parent(s) or legal guardian(s) and by the patient, if capable
* Prepubertal stage
* Good health with the exception of asthma
* History of asthma for at least 6 months
* Currently using rescue medication only

Main Exclusion Criteria:

* Childbearing potential (beyond menarche)
* Concurrent diseases or conditions which may subsequently affect growth
* COPD or relevant lung diseases causing alternating impairment in lung function
* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* History of life-threatening asthma
* Current smoking

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28
Dates: Start 2005-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
growth velocity of the right lower leg as measured by knemometry.

SECONDARY OUTCOMES:
HPA-axis function
weight and height
lung function from spirometry
asthma symptom score, use of rescue medication from diary
adverse events
vital signs, including blood pressure, pulse rate
physical examination
laboratory investigation.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Altana Pharma/Nycomed, Kolding, Denmark

REFERENCES:
- See also: BY9010-MI-208-RDS-2007-04-11.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4528&filename=BY9010-MI-208-RDS-2007-04-11.pdf